CLINICAL TRIAL: NCT02599714
Title: A Phase I/II Multicenter Study of the Combination of AZD2014 and Palbociclib on a Background of Hormonal Therapy in Patients With Locally Advanced/Metastatic Estrogen Receptor Positive Breast Cancer Comprising a Safety, Pharmacokinetic and Preliminary Efficacy Evaluation Followed by a Randomized, Double-Blind, Placebo-controlled, Parallel Group Extension (PASTOR).
Brief Title: Study of AZD2014 and Palbociclib in Patients With Estrogen Receptor Positive (ER+) Metastatic Breast Cancer
Acronym: PASTOR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2270C00020; 264477 (Other: Parexel International Corporation); 2015-003320-30 (EudraCT Number)
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Advanced and Metastatic Breast Cancer
Keywords: AZD2014; Palbociclib; Fulvestrant; Hormonal Therapy; Estrogen Receptor Positive; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — vistusertib; palbociclib; Fulvestrant

STUDY DESIGN:
Masking Description: Study was originally designed as randomized and double blinded. Currently (CSP v.8.0 of 14-Dec-2021) no masking and no randomization is planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Triplet Combination (Dose Finding) (Experimental): Phase 1 triplet dose finding phase in 3-6 patients per cohort - approximately 30 patients depending on emerging data to determine the maximum tolerated dose (MTD) of the triplet.
  Interventions: Drug: AZD2014; Drug: Palbociclib; Drug: Fulvestrant
- Triplet Combination (Dose Expansion) (Experimental): Additional patients will be enrolled at the dose determined in Part A.
  Interventions: Drug: AZD2014; Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: AZD2014 — The triplet combination will be comprised of AZD2014 + palbociclib + fulvestrant.
  Other Names: vistusertib
Drug: Palbociclib — cyclin dependent kinase inhibitor
  Other Names: Ibrance; PD-0332991
Drug: Fulvestrant — Fulvestrant hormonal therapy as background
  Other Names: Faslodex

SUMMARY:
This dose finding/extension study was designed originally to consist of three parts: Part A was intended to identify the MTD of the AZD2014/ palbociclib combination on a background of fulvestrant (referred to as the triplet) in postmenopausal women with locally advanced/ metastatic estrogen receptor positive (ER+) breast cancer. Part B was to further characterize safety, tolerability, PK, and preliminary efficacy in single-arm dose expansion groups. Part C was to be a Phase 2, randomized, double-blind, extension comparing the triplet and doublet combinations. Part C was deleted from the protocol and was not performed.

DETAILED DESCRIPTION:
This dose finding/extension study was designed originally to consist of three parts:

Part A is a Phase 1 triplet-dose finding investigation in 3-6 patients per cohort to determine the maximum tolerated dose (MTD) of the triplet.

Part B is a single arm expansion in approximately 27 patients evaluable for response to define the recommended Phase 2 dose (RP2D).

Part C was intended to investigate the efficacy of the triplet combination at the RP2D in a randomized, double-blind, placebo-controlled, stratified, parallel group extension. Part C was intended to include ER+, locally advanced and/or metastatic breast cancer patients who have progressed following prior non-steroidal aromatase inhibitor (NSAI) endocrine therapy. Patients in Part C were to be randomized to receive either the triplet combination (AZD2014 + palbociclib + fulvestrant) or the doublet (matching AZD2014 placebo + palbociclib + fulvestrant). Patients were to be stratified according to hormone sensitivity, presence of visceral metastases, and prior CDK inhibitor treatment. Part C would have been conducted if indicated by the emerging data.

ELIGIBILITY:
Inclusion:

1. Signed and dated written informed consent prior to any mandatory study specific procedures, sampling and analyses.
2. Signed and dated written informed consent for tumour biopsies. If the tumour is found not to be safely accessible the biopsy will not be taken. Accessible lesions are defined as those which are biopsiable and amenable to repeat biopsy, unless clinically contraindicated. In this case the patient will remain in the study and there will be no penalty or loss of benefit to the patient and they will not be excluded from other aspects of the study.
3. Postmenopausal women aged ≥ 18 years
4. Negative pregnancy test prior to dosing and willing to use a highly effective method of contraception for the duration of the study and for 90 days after the last dose of IP if they are under 50 unless they have medically confirmed irreversible premature ovarian failure, bilateral oophorectomy, bilateral salpinectomy, or complete or partial hysterectomy.

   Highly effective methods of contraception are:

   • Use of oral, injected or implanted hormonal methods of contraception which inhibit ovulation, either estrogen and progestogen containing intravaginal, transdermal) or only progesterone containing (oral, injectable, implantable)

   • Placement of an intrauterine device (IUD or intrauterine system (IUS)

   • True abstinence
   * Bilateral tubal ligation
   * Vasectomised partner
5. World Health Organisation/Eastern Cooperative Oncology Group (ECOG) performance status of patient is 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks.
6. Histologically or cytologically proven diagnosis of breast cancer with evidence of locally advanced or metastatic disease, not amenable to resection or radiation therapy with curative intent.
7. Documentation of estrogen receptor positive (ER+) breast cancer based on most recent tumour biopsy (unless bone-only disease).
8. Documented human epidermal growth factor receptor 2 negative (HER2-) tumor on most recent tumor biopsy.
9. Where regionally permitted, all patients must agree to provide if available a formalin-fixed paraffin embedded (FFPE) tissue biopsy sample taken at the time of presentation with recurrent or metastatic disease.
10. At least one lesion (measurable and/or non measurable) that can be accurately assessed at baseline with computerised tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements.
11. Meet the following study part specific criteria related to previous therapy for breast cancer:

For Part A: Postmenopausal patient suitable for fulvestrant. Patient is allowed to have a maximum of 3 prior lines of chemotherapy. Previous treatment with CDK4/6 inhibitors is allowed

For Part B: Postmenopausal patient with locally advanced or metastatic ER+ve breast cancer and refractory to AIs defined as:

* Disease recurrence while on, or within 12 months of end of adjuvant treatment with letrozole, anastrozole, or exemestane, or
* Disease progression while on, or within one month of end of letrozole, anastrozole or exemestane treatment for locally advanced or metastatic breast cancer

  * Letrozole or anastrozole do not have to be the last treatment prior to randomization.
  * Patients who received one prior chemotherapy line for advanced/metastatic breast cancer are allowed.

Previous treatment with fulvestrant (or letrozole) is allowed. Other prior anticancer therapy (e.g. tamoxifen) are also allowed.

For inclusion in the optional research component:

1. Genetic research: Provision of signed and dated written consent for genetic research sampling and analyses. If a patient declines to participate in genetic component of the study, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study described in this Clinical Study Protocol, so long as they consent to the main study.

Exclusion:

1. Prior chemotherapy, biological therapy, radiation therapy, or immunotherapy, androgens, thalidomide, other anticancer agents, investigational drug or corticosteroids within 14 days. Patients who received prior radiotherapy to >= 25% of bone marrow are not eligible independent of when it was received. Patients is not eligible if there are unresolved toxicities from prior therapy > CTCAE grade 1 at the start of study treatment with the exception of alopecia.
2. Exposure to potent or moderate inhibitors or inducers of CYP3A4/5, Pgp (MDR1) or BCRP within stated washout periods.
3. Exposure to sensitive or narrow therapeutic range substrates of drug transporters OATP1B1, OATP1B3, MATE1 and MATE2K within wash-out period (5 x elimination half-life).

4 Exposure to proton pump inhibitors within wash-out period (5 x elimination half-life).

5. Previous AZD2014, AZD8055 or other dual mTORC1/2 inhibitor

* In Part B only: Prior treatment with CDK4/6, or everolimus or any PI3K-mTOR pathway

  6. Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease. Patients with a history of CNS metastases or cord compression are eligible if definitively treated and clinically stable and off anticonvulsants and steroids for at least 4 weeks. Patients are not eligible if there is spinal cord compression and/or brain metastases, unless asymptomatic or treated and stable and off steroids for at least 4 weeks.

  7. Evidence of severe or uncontrolled systemic diseases such as:

  • Severe hepatic impairment

  • Interstitial lung disease (bilateral, diffuse, parenchymal lung disease)
  * Current unstable or uncompensated respiratory or cardiac conditions
  * Uncontrolled hypertension
  * Active bleeding diatheses
  * Any active infection

    8. Other malignancy within 3 years, except adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix

    9. Experienced any of the following currently or in the last 12 months:
  * Coronary/peripheral artery bypass graft
  * Angioplasty
  * Vascular stent
  * Myocardial infarction
  * Angina pectoris
  * Congestive heart failure NYHA Grade ≥ 2
  * Ventricular arrhythmias requiring continuous therapy
  * Supraventricular arrhythmias including atrial fibrillation of any grade
  * Symptomatic pulmonary embolism
  * Haemorrhagic or thrombotic stroke

    10. Abnormal ECHO or MUGA at baseline (LVEF <50%).

    11. Mean resting QTc >470 msec, family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes within 12 months.

    12. Clinically important abnormalities in rhythm, conduction or morphology of resting ECG.

    13. Hepatitis B (HBV), Hepatitis C (HCV) or Human Immunodeficiency virus (HIV).

    14. Concomitant medications known to predispose to Torsade de Pointes, or factors that increase the risk of QT prolongation or risk of arrhythmic events such as:
  * Heart failure
  * Hypokalaemia
  * Congenital long QT syndrome
  * Family history of long QT syndrome
  * Family history of unexplained sudden death under 40 years-of-age

    15. Inadequate bone marrow reserve or organ function as demonstrated by:
  * ANC <1.5 x 10^9/L.
  * In Part A only - Cohorts of patients with specific baseline ANC range to be enrolled defined as follows: I) Low ANC patients: between 1.5 x 10^9/L and 3.0 x 10^9/L; ii) High ANC patients > 3.0 x 10^9/L.
  * Platelets <100 x 10^9/L
  * Haemoglobin <90 g/L
  * ALT >2.5 x ULN or > 5 x ULN in the presence of liver mets.
  * AST >2.5 x ULN or > 5 x ULN in the presence of liver mets.
  * Total bilirubin >1.5 x ULN. Total bilirubin >3 x ULN in patients with documented Gilbert's Syndrome.
  * Serum creatinine >1.5 x ULN concurrent with creatinine clearance ≤50 mL/min.

    16. Pre-existing renal disease including glomerulonephritis, nephritic syndrome, Fanconi Syndrome or Renal tubular acidosis.

    17. Refractory nausea/vomiting, chronic GI diseases, inability to swallow the product or previous significant bowel resection.

    18. Hypersensitivity to excipients of AZD2014, Palbociclib or Fulvestrant or drugs with a similar structure.

    19. Diabetes Type I or uncontrolled Type II, as defined in WHO 2006 (fasting serum glucose of > 7.0 mmol/L [126 mg/dL]).

    20. Patient with advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term including patients with massive uncontrolled effusions (pleural, pericardial, peritoneal), pulmonary lymphangitis, and over 50% of liver involvement in metastases.

    21. Prior hematopoietic stem cell or bone marrow transplant.

    22. Regular coumadin therapy. Low-molecular-weight heparin therapy or oral Factor Xa antagonists are allowed.

    23. Known abnormalities in coagulation, e.g. bleeding diathesis.

    24. Hematopoietic growth factors (such as erythropoietin, granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony stimulating factor [GM-CSF]) within 2 weeks prior. Primary prophylactic use of G-CSF is not permitted.

    25. Other severe acute or chronic psychiatric condition that may increase the risks associated with study participation.

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2015-12-07 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Parts A and B: Number of adverse events experienced by patients | Approximately 16 months
  Safety and tolerability assessed through the incidence of adverse events.

SECONDARY OUTCOMES:
Part B: Progression Free Survival (PFS) | Assessed every 8 weeks for approximately 16 months
  PFS assessed through change in tumour size (as well as assessment of non-target lesions and appearance of any new lesions) according to RECIST 1.1 criteria by Investigator assessment.
Parts A and B: Best Objective Response (BOR) | Assessed every 8 weeks for approximately 16 months
  BOR assessed according to RECIST 1.1 criteria by Investigator assessment.
Parts A and B: Objective Response Rate (ORR) | Assessed every 8 weeks for approximately 16 months
  ORR assessed through the number of patients who achieve a disease response (i.e. complete response or partial response) according to RECIST 1.1 criteria
Part B: Duration of Response (DoR) | Assessed every 8 weeks for approximately 16 months
  DoR assessed as the time between disease response being achieved and progressive disease as assessed by RECIST 1.1 criteria or end of life (in the absence of progression)
Part B: Overall Survival (OS) | Approximately 24 months
  The time from start of treatment until end of life from any cause.
Part A: Peak plasma concentrations (Cmax) of AZD2014 and palbociclib following single dose | Samples for single dose PK will be collected at prespecified time points up to 12 hours following dosing.
  Venous blood samples for determination of concentrations of AZD2014 and palbociclib in plasma will be collected.
Parts A and B: Peak plasma concentrations (Cmax) of AZD2014 and palbociclib following multiple doses | Samples will be collected at prespecified time points up to 12 hours following dosing.
  Venous blood samples (2 mL for each drug) for determination of concentrations of AZD2014 and palbociclib in plasma will be collected.
Parts A and B: Change from baseline in biomarker H-score | 16 months
  For those subjects with paired tumour biopsies the pharmacodynamic markers will be assessed by immunohistochemistry.
Time to reach peak plasma concentrations (tmax) for AZD 2014 and palbociclib. | Samples will be collected at prespecified time points up to 12 hours following dosing.
  The plasma concentrations of AZD2014 and palbociclib will be determined. Tmax is the time required after administration for the drug to reach its peak plasma concentration.
Area under the plasma concentration-time curve from zero to 12 hours (AUC 0-12) for AZD 2014 and palbociclib. | Samples will be collected at prespecified time points up to 12 hours following dosing.
  The plasma concentrations of AZD2014 and palbociclib will be determined. Area under the curve is the integral of the concentration-time curve. The area under the plasma drug concentration-time curve (AUC) reflects the actual body exposure to drug after administration. The area under the curve is dependent on the rate of elimination of the drug from the body and the dose administered.
Area under the plasma concentration-time curve from zero to 24 hours (AUC 0-24) for AZD 2014 and palbociclib. | Samples will be collected at prespecified time points up to 24 hours following dosing.
  The plasma concentrations of AZD2014 and palbociclib will be determined. Area under the curve is the integral of the concentration-time curve. The area under the plasma drug concentration-time curve (AUC) reflects the actual body exposure to drug after administration. The area under the curve is dependent on the rate of elimination of the drug from the body and the dose administered.
Area under the plasma concentration-time curve from zero to the last measurable concentration (AUC 0-t) for AZD 2014 and palbociclib. | Samples will be collected at prespecified time points up to 9 days following dosing.
  The plasma concentrations of AZD2014 and palbociclib will be determined. Area under the curve is the integral of the concentration-time curve. The area under the plasma drug concentration-time curve (AUC) reflects the actual body exposure to drug after administration. The area under the curve is dependent on the rate of elimination of the drug from the body and the dose administered.
Area under the plasma concentration-time curve from zero to infinity (AUC 0-∞) for AZD 2014 and palbociclib. | Samples will be collected at prespecified time points up to 9 days following dosing.
  The plasma concentrations of AZD2014 and palbociclib will be determined. Area under the curve is the integral of the concentration-time curve. The area under the plasma drug concentration-time curve (AUC) reflects the actual body exposure to drug after administration. The area under the curve is dependent on the rate of elimination of the drug from the body and the dose administered.
Terminal elimination rate constant (λz) for AZD 2014 and palbociclib. | Samples will be collected at prespecified time points up to 9 days following dosing.
  The plasma concentrations of AZD2014 and palbociclib will be determined. The elimination rate constant is the rate at which drug is cleared from the body assuming first-order elimination
Terminal plasma half-life (t1/2λz) for AZD 2014 and palbociclib. | Samples will be collected at prespecified time points up to 9 days following dosing.
  The plasma concentrations of AZD2014 and palbociclib will be determined. The terminal plasma half-life is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium.

CONTACTS AND LOCATIONS:
Overall Officials: Anja Wiliams, Principal Investigator — Sarah Cannon Research Institute UK
Locations (7):
- United States (5):
  - Research Site, Encinitas, California
  - Research Site, Sarasota, Florida
  - Research Site, Detroit, Michigan
  - Research Site, Nashville, Tennessee
  - Research Site, Milwaukee, Wisconsin
- United Kingdom (2):
  - Research Site, Liverpool
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2270C00020&attachmentIdentifier=7769c909-c2e1-4547-9b6c-491f834d0089&fileName=d2270c00020-study-synopsis_Redacted.pdf&versionIdentifier=